CLINICAL TRIAL: NCT00638131
Title: Effect of Bosentan on Systemic and Renal Inflammatory Markers in Patients With Diabetic Nephropathy on Angiotensin II Receptor Blockers
Brief Title: Bosentan Use in Patients With Diabetic Nephropathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: problem of recruitment
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BOS-ND-2007
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2010-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Bosentan 62.5mg bid x4 weeks; up-titrated to 125mg bid x12 weeks;
  Interventions: Drug: bosentan
- 2 (Placebo Comparator): placebo given bid same as experimental arm;
  Interventions: Drug: bosentan

INTERVENTIONS:
Drug: bosentan — 62.5mg bid x4 weeks, up-titrate to 125mg bid x12 weeks
  Other Names: Tracleer

SUMMARY:
There is little doubt of the necessity for further improvement in the prevention and therapy of end-stage renal disease. Despite the success of ARB in treating diabetic nephropathy, not all patients obtain satisfactory control of blood pressure, albuminuria and decline in renal function. Experimental data have provided us with a rationale for the potential added benefits of ET receptor blockade to the AII inhibition in diabetic renal protection. Considering the nephroprotective effect of bosentan in diabetic rats, clinical studies are warranted to assess whether ET receptor antagonism has additive renoprotective effects on top of AII inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years of age with a body weight of ≥ 40 kg;
* For female patients, only non-pregnant women who are surgically sterile, postmenopausal or have documented infertility (over 50 years of age and amenorrheic for at least 1 year), or those of childbearing potential using intrauterine devices (IUDs);
* Patients diagnosed Type 2 diabetes with overt nephropathy (urinary albumin excretion ≥ 300mg/24h);
* Patients on current treatment with angiotensin II receptor blockers for ≥ 3 months;
* Patients stable for at least 3 months prior to screening (no change in medications for diabetic nephropathy);
* Provide written informed consent;

Exclusion Criteria:

* Patients with a history of pulmonary chronic obstructive disease, cardiac failure or coronary artery disease;
* Patients with documented cancers, acute infections or chronic inflammatory diseases;
* Patients who are pregnant or breast-feeding;
* Patients with known hepatic disorders or AST and ∕or ALT upper than normal limit;
* Patients with hemoglobin or hematocrit that is ≥ 30% below the normal range (patients with secondary polycythemia are permitted);
* Patients with systolic blood pressure < 110mm Hg;
* Patients with plasmatic albumin level < 30g/L;
* Patients with a documented creatinine clearance ≤ 60ml/min;
* Patients on anticoagulants or anti-inflammatory drugs, including cyclooxygenase inhibitors, AINS, prednisone and immunosuppressive drugs, platelet aggregation inhibitors, except low dose aspirin, ACE inhibitors, antidiabetic agents (rosiglitazone, pioglitazone) and antioxidants (vitamin E)(except statins or low-dose aspirin ≤ 80mg/day);
* Patients on treatment or planned treatment with another investigational drug;
* Patients who are receiving an endothelin receptor antagonist, phosphodiesterase type 5 inhibitor, or with a prostanoid (excluding acute administration during a catheterization procedure to test vascular reactivity) within 2 months of inclusion;
* Patients who are receiving calcineurin-inhibitors (i.e., cyclosporine A and tacrolimus), fluconazole, glibenclamide (glyburide) at inclusion or are expected to receive any of these drugs during the study;
* Patients with a known hypersensitivity to bosentan or any of the excipients;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
change from baseline to week 16 in renal inflammation. The following urinary inflammatory/oxidative stress parameters will be measured: - TNF | 16 weeks

SECONDARY OUTCOMES:
change from baseline to week 16 in renal functioning. The following renal function parameter will be measured: - 24h UAE; | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maryse Courteau, MD, Principal Investigator — CHUM
Locations (1):
- CHUM, Montreal, Quebec, Canada